CLINICAL TRIAL: NCT03040921
Title: Uterine Transposition: Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Erasto Gaertner (Other)
Responsible Party: Principal Investigator, Reitan Ribeiro, MD, Hospital Erasto Gaertner
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HEG01
Record Dates: First submitted 2017-01-14; First posted 2017-02-02 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Complications; Intraoperative Complications; Tissue Damage; Ovarian Failure; Uterus Disorder
MeSH Terms: conditions — Postoperative Complications; Intraoperative Complications; Uterine Diseases

STUDY DESIGN:
Intervention Model Description: Recruitment completed. Final data collection in April/2020.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uterine Transposition (Experimental): Patients submitted to uterine transposition.
  Interventions: Procedure: Uterine transposition.

INTERVENTIONS:
Procedure: Uterine transposition. — Surgical transposition of the uterus to the upper abdomen. After the end of radiotherapy, rectosigmoidectomy is performed and the uterus is repositioned into the pelvis.

SUMMARY:
This prospective nonrandomized multicenter phase I study, will evaluate the feasibility of performing uterine transposition before chemoradiation for rectal cancer and uterine reimplantation after the treatment.

DETAILED DESCRIPTION:
Patients with pelvic cancer frequently require radiotherapy, which causes infertility even at low doses. Oocytes are highly sensitive to radiation, as a dose of 2 Gy is able to destroy up to 50% of the oocyte population.

Pelvic radiotherapy with fertility preservation is not yet available for women with pelvic tumors. In such cases, the only options are egg and/or embryo freezing and ovarian transposition (OT), which might preserve reproductive and hormonal function, respectively. While ovarian tissue cryopreservation and transplantation are possible, they are still experimental.

Uterine and adnexal transposition (UT) to the upper abdomen before radiotherapy might protect these organs, and the later repositioning of the uterus into the pelvis after radiotherapy might allow the patients to experience a normal pregnancy.

Methods:

Patients with pelvic cancer who will need pelvic radiation will be offered the possibility to performed the uterine transposition before the radiation therapy and after the treatment the uterus will be replaced in it's natural position. The study period is 2 years or 10 patients, that happens first.

The suggested treatment consisted of oocyte or embryos vitrification or before the uterine transposition, but this is not mandatory.

Patient preparation, equipment and trocars placement will be performed as usual for pelvis procedures and retroperitoneal dissection. The following provides each step of the surgical procedure: sealing and section of the round ligament; opening of the broad ligament; dissection of the vesicovaginal space; sealing and section of the uterine vessels at the level of the cervix; sealing and sectioning of the pericervical vessels and uterosacral ligaments; Section of the vagina. Closure of the vagina with absorbable sutures; dissection of the infundibulopelvic (IP) ligaments up to their intersection with the iliac vessels; separation of the terminal ileum, right, sigmoid and descending colon from the retroperitoneal space to allow dissection of the gonadal vessels up to their origin; transposition of the uterus to the upper abdomen, and repositioning of the colon and ileum bellow the arch formed by the uterus, adnexa and the corresponding vessels; fixation of the round ligaments and gonadal vessels to the upper abdomen by means of a transparietal suture to avoid herniation or by moving them into the pelvis; draining the pneumoperitoneum and placement of transabdominal sutures at the site; fixation of the cervix to the umbilical incision to allow for menstruation from the navel; and visual inspection of the cervix, which indicates the end of the surgical procedure. The adnexa should not be contacted at any time during surgery.

Postoperative care will be performed as for major procedures in gynecology. Visual inspection of the cervix will be performed twice per day, and uterine perfusion was assessed every 2 days by Doppler ultrasound of the ovarian vessels. The patient is discharged 2-4 days after surgery if no complications occur. Three-dimensional radiotherapy or Intensity-Modulated Radiation Therapy following the standard treatment for the disease will start 10 to 14 days later. Chemotherapy may be used, also following the usual treatment. Chemotherapy and radiotherapy protocols must follow the standard treatment of the disease, no adaptations are accepted.

Five weeks after the end of radiotherapy, in rectal cancer cases, rectosigmoidectomy with total mesorectal excision (TME) and repositioning of the uterus will be performed. Patients with other tumors that do not need surgery as part of its treatment, the uterine repositioning will be performed 7 - 30 days after the end of the treatment.

The repositioning procedures is performed as follows: First, the cervix is separated from the navel, and the first trocar is inserted. Second, adhesions are removed, and the uterus and adnexa are repositioned into the pelvis. Rectosigmoidectomy with laparoscopic TME then followed the usual technique., Chromotubation is performed at the end of the procedure to demonstrate tubal patency. Patients without complications are expected to be discharged 2 - 4 days after surgery.

Seven days after surgery, cervical inspection is performed. Image exams will be performed as clinically indicated in the postoperative period. Clinical evaluation with pelvic examination will be performed every week for 4 weeks, then every months for 6 months and after that every 3 months for 2 years. Complications form will be filled in all clinical evaluations. Every 3 months, quality of life protocols will be applied. Abdominal and pelvic Magnetic resonance will be performed 1, 6 and 12 months after the surgery. Transvaginal ultrasound will be performed 2, 4 and 6 months after the surgery. Hormonal evaluation will be performed every 3 months. Tumor follow-up will be performed according to the institution protocols. It is recommend to the patients to wait for 1 year before trying pregnancy.

Reports concerning safety will be presented every 6 months to the local Ethics Committee. No uterine necrosis is expected and in case of 2 uterine necrosis, the study will be stoped. Up to two local recurrences in the study period are accepted, but in case of a third recurrence, the study will be stoped. All complication will be reviewed by the local board and the study will be under permanent evaluation. Every 6 months the local board will provide a report allowing the study to continue or not.

ELIGIBILITY:
Inclusion Criteria:

* Women with pelvic cancer and indication for pelvic radiation therapy who have fertility sparing desire.

Exclusion Criteria:

* Previously documented infertility, ovarian failure or gynecologic cancer.
* More than 40 yo.
* Previous oophorectomy
* Tumor infiltrating uterus or adnexes
* Presence of peritoneal metastasis
* Presence of systemic metastasis
* Previous retroperitoneal radiotherapy
* Retroperitoneal radiotherapy planned

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Uterine preservation after transposition to the upper abdomen and replacement in the pelvis | 6 months
  The preservation of the uterus with normal endometrium confirmed by ultra-sound, after the surgery to place it in the upper abdomen and after replacing the uterus back to its normal position.

SECONDARY OUTCOMES:
Morbidity | 6 months
  Intraoperative and postoperative complications
Cancer recurrence | Through study completion, an average of 2 years
  Local and distant recurrences

CONTACTS AND LOCATIONS:
Overall Officials: Reitan Ribeiro, MD, Principal Investigator — Erasto Gaertner Hospital
Locations (1):
- Erasto Gaertner Hospital, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No
Hospital Ethics Committee did not approve individual participant data sharing. Recruitment completed. Final data collection in April/2020.

REFERENCES:
- See also: Erasto Gaertner Hospital webpage — https://erastogaertner.com.br/